CLINICAL TRIAL: NCT01912885
Title: Comparison of Posterior Tibial Nerve Electrical Stimulation Protocols for Overactive Bladder Syndrome: Randomized Blind Clinical Trial
Brief Title: Comparison of Posterior Tibial Nerve Electrical Stimulation Protocols for Overactive Bladder Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MunickP
Record Dates: First submitted 2013-06-05; First posted 2013-07-31 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2017-12

CONDITIONS: Overactive Bladder Syndrome

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group TENS 0-1 (Placebo Comparator): Electrodes will be fixated to one leg and sessions will be held once a week.
  Interventions: Device: TENS 0-1
- Group TENS 1-1 (Experimental): Electrical stimulation of the posterior tibial nerve of one leg once a week.
  Interventions: Device: TENS 1-1
- Group TENS 1-2 (Experimental): Electrical stimulation of the posterior tibial nerve of one leg twice a week.
  Interventions: Device: TENS 1-2
- Group TENS 2-1 (Experimental): Electrical stimulation of the posterior tibial nerve of two legs once a week.
  Interventions: Device: TENS 2-1
- Group TENS 2-2 (Experimental): Electrical stimulation of the posterior tibial nerve of two legs twice a week.
  Interventions: Device: TENS 2-2

INTERVENTIONS:
Device: TENS 1-1 — Electrical stimulation using Transcutaneous Electrical Nerve Stimulation on one leg once a week.
  Arms: Group TENS 1-1
Device: TENS 1-2 — Electrical stimulation using Transcutaneous Electrical Nerve Stimulation on one leg twice a week.
  Arms: Group TENS 1-2
Device: TENS 2-1 — Electrical stimulation using Transcutaneous Electrical Nerve Stimulation on two legs once a week.
  Arms: Group TENS 2-1
Device: TENS 2-2 — Electrical stimulation using Transcutaneous Electrical Nerve Stimulation on two legs twice a week.
  Arms: Group TENS 2-2
Device: TENS 0-1 — Placebo: application os electrodes of Transcutaneous Electrical Nerve Stimulation on one leg once a week, without turning on the device.
  Arms: Group TENS 0-1

SUMMARY:
INTRODUCTION: Overactive bladder syndrome is defined by The International Continence Society as urgency, with or without incontinence, usually with increased urinary frequency and nocturia. It is difficult to estimate the prevalence of this syndrome because many patients do not seek medical help, despite considerable negative impact on quality of life. Lower urinary tract dysfunctions can be treated using electrical stimulation of the posterior tibial nerve. This therapy is conservative, effective, inexpensive and promotes high adhesion to treatment. It has good results, decreasing symptoms of urgency, urge-incontinence, urinary frequency and nocturia . Due to lack of consensus on the parameters of this technique, further research is necessary. OBJECTIVE: To compare the effectiveness of protocols for the electrical stimulation of the posterior tibial nerve for treatment of non-neurogenic overactive bladder. METHODS: The study was a blind randomized clinical trial. The study will accept up to 145 women with overactive bladder diagnosis for at least six months prior to the beginning of the study. The subjects will be divided into five groups: group TENS 0-1 (placebo group), group TENS 1-1 (electrical stimulation of one leg once a week), group TENS 1-2 (electrical stimulation of one leg twice a week), group TENS 2-1 (electrical stimulation of two legs one a week) and group TENS 2-2 (electrical stimulation of two legs twice a week). Physical evaluation will be done at the beginning and at the end of the treatment. Evaluation will be done using the King "s Health Questionnaire, the International Consultation Incontinence Questionnaire - Short Form, the Overactive Bladder Questionnaire, a three day urinary diary and a table for follow-up treatment.

DETAILED DESCRIPTION:
Participants will be recruited from Urogynecology Physical Therapy Outpatient Clinic of a university hospital and randomly assigned using website www.randomization.com and distributed into five groups considering the sites of application and frequency of attendanc, listed above.

Data will be collected by the investigator using interview and physical examination and will be safely stored in computer.

For this study, in terms of urinary frequency, the standard deviation was estimated at 3.25 episodes of urinary urgency (SD=3.25). With 80% power and 95% confidence, the sample size calculation was 25 women in each group, plus a possible sample loss of around 20%, resulting in a sample size of 29 women per group, for a total of 145 patients in the study.

The chi-square test was used to assess whether there was an association between sample description variables and treatments. The analysis of variance F-test was used to assess whether there were differences in the numerical descriptive variables between treatment groups. The nonparametric Kruskal-Wallis test was used to compare treatments in terms of the difference between before and after for each quality of life and voiding diary variables. If there was statistical significance, the Dunn multiple comparison test was performed, with p-values of less than 0.05 considered significant. The analysis of variance model with repeated measures was used to compare data from the specific voiding diary according to the treatment groups and sessions. Significant comparisons were evaluated with Tukey post-hoc test. To approximate data to the normality, a 1/log (variable+1) transformation was done. For the follow up analysis, it was used the ANOVA three ways, with Holm Sidak post-hoc test for comparison of scores. All the statistical tests developed were based on a significance of 5%, i.e., the null hypothesis was rejected when the p-value was less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Women with 18 years of age or more;
* Cognitive level adequate for understanding orientations during treatment;
* Clinical diagnosis of overactive bladder syndrome for at least six months prior to the study.

Exclusion Criteria:

* Pregnant women or women who wish to get pregnant;
* Neurological disease;
* Urinary infection;
* Nephrolithiasis;
* Stress urinary incontinence;
* Mixed urinary incontinence;
* Women in pharmacological treatment for overactive bladder syndrome;
* Women undergoing hormone replacement therapy in the last six months;
* Peripheral neuropathy;
* Cystocele stage two or higher.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2013-10-09 (Actual); Primary Completion 2014-08-25 (Actual); Study Completion 2014-09-25 (Actual)

PRIMARY OUTCOMES:
Change in urinary frequence in 12 sessions. | The patients fill in a bladder diary of 3 days running. One bladder diary starting in the first session and the last one to end in the last session.
  Number of micturitions per day.

SECONDARY OUTCOMES:
Change in Nocturia in 12 sessions. | The patients fill in a bladder diary of 3 days running. One bladder diary starting in the first session and the last one to end in the last session.
  Number of micturitions per night, interrupting sleep.
Change in urinary urgence in 12 sessions. | The patients fill in a bladder diary of 3 days running. One bladder diary starting in the first session and the last one to end in the last session.
  Number of urgent micturitions per day.
Change in urinary urge-incontinence in 12 sessions. | The patients fill in a bladder diary of 3 days running. One bladder diary starting in the first session and the last one to end in the last session.
  Number of leaks per day.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth AG Ferreira, PhD, Study Director — Faculty of Medicine, University of São Paulo, São Paulo, Brazil
Locations (1):
- Gynecology Ambulatory of the General Hospital of the Faculty of Medicine of the University of Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Pierre ML, Friso B, Casarotto RA, Haddad JM, Baracat EC, Ferreira EAG. Comparison of transcutaneous electrical tibial nerve stimulation for the treatment of overactive bladder: a multi-arm randomized controlled trial with blinded assessment. Clinics (Sao Paulo). 2021 Aug 16;76:e3039. doi: 10.6061/clinics/2021/e3039. eCollection 2021. PMID 34406271